CLINICAL TRIAL: NCT02386397
Title: Activity of Regorafenib in Combination With Modified Gemcitabine - Oxaliplatin Chemotherapy (mGEMOX) in Patients With Advanced Biliary Tract Cancer (BTC): A Phase Ib-II Trial (BREGO)
Brief Title: Activity of Regorafenib in Combination With Chemotherapy in Patients With Advanced Biliary Tract Cancer
Acronym: BREGO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICM2013/09
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2017-08

CONDITIONS: Digestive Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — regorafenib; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Regorafenib: X mg/d, PO, from day 1 to day 14; day 15 to day 20: off-treatment mGEMOX: infusion on days 1 and 8
  * Gemcitabine 900 mg/m² IV in 30 minutes
  * Oxaliplatin 80 mg/m² IV in 120 minutes immediately after Gemcitabine
  Interventions: Drug: Regorafenib; Drug: GEMOX
- Standard treatment (Other): mGEMOX: infusion on days 1 and 8
  * Gemcitabine 900 mg/m² IV in 30 minutes
  * Oxaliplatin 80 mg/m² IV in 120 minutes immediately after Gemcitabine
  Interventions: Drug: GEMOX

INTERVENTIONS:
Drug: Regorafenib — Regorafenib: X mg/d, PO, from day 1 to day 14; day 15 to day 20: off-treatment
  Other Names: Gemcitabin; Oxaliplatin
  Arms: Treatment
Drug: GEMOX — mGEMOX: infusion on days 1 and 8: Gemcitabine 900 mg/m² IV in 30 minutes Oxaliplatin 80 mg/m² IV in 120 minutes immediately after Gemcitabine
  Other Names: Gemcitabine; Oxaliplatin

SUMMARY:
This study is to determine the Regorafenib Dose (RD) for the phase II trial of Regorafenib administered in combination with mGEMOX in patients with advanced biliary tract cancer.

DETAILED DESCRIPTION:
Regorafenib (BAY 73-4506) was assessed in metastatic colorectal cancer in the phase III randomized CORRECT trial. 760 metastatic colorectal cancer patients were recruited after the failure of all standard therapies.

Given the promising efficacy and favorable tolerability profile of mGEMOX and the potential benefits of targeting the VEGF and Ras/Raf pathway, we propose to assess the combination of Regorafenib with mGEMOX in advanced digestive cancer.

This study is to determine the Regorafenib Dose (RD) for the phase II trial of Regorafenib administered in combination with mGEMOX in patients with advanced biliary tract cancer.

The phase I study of Regorafenib in advanced colorectal cancer showed a pronounced interindividual variability of drug exposition. Furthermore, the CORRECT study shows a large pharmacological variability of plasma concentration for Regorafenib and its metabolites. In this study, we propose to explore the pharmacological variability and his potential heritability by the therapeutic drug monitoring of Regorafenib. The objective is to understand and to control the pharmacological variability of Regorafenib and finally to predict the therapeutic response or the toxicity, especially in a population of patients with biliary tract cancer.

In addition, we will complete this study by exploring the gene variants of drug metabolism. The genes are POR (P450 OxidoReductase,) NR1I2 (Nuclear Receptor subfamily 1, group I, member 2) and a part of the regulatory sequences of CYP3A4.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the biliary tract
* Metastatic disease with no curative surgery option or metastatic recurrence after resection.
* Only for phase II: At least one measurable lesion in a non-irradiated area according to Response Evaluation Criteria in Solid Tumors
* No biliary obstruction.
* Age between 18 and 75 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy higher than 3 months.
* No prior chemotherapy for advanced disease. Previous adjuvant chemotherapy including Gemcitabine and/or platinum based is allowed if completed at least 6 months previously and relapsing after completion of the last dose.
* Total bilirubin ≤ 2.5 times the upper limit of the normal range. Patients with jaundice or evidence of bile duct obstruction, in whom the biliary tree can be decompressed by endoscopic or percutaneous endoprothesis (at least 15 days before inclusion) with subsequent reduction in total bilirubin ≤ 3 ULN, will be eligible for the study.
* Aminotransferases (AST, ALT) ≤ 2.5 ULN (≤ 5 ULN in case of diffuse hepatic involvement), INR < 1.5 (following vitamin K1 injection in patients with current or recent history of jaundice or bile duct obstruction), serum creatinine clearance calculated > 50 mL/min/1.73m² according to the Modification of Diet in Renal Disease (MDRD) formula, neutrophils ≥ 1.5.109/L, platelets ≥ 100.109/L, hemoglobin ≥ 9 g/dL (red blood cell transfusion is allowed if needed).
* Signed informed consent obtained before any study specific procedures.
* Patients must be affiliated to a Social Security System.

Exclusion Criteria:

* Known central nervous system metastases.
* Known history of human immunodeficiency virus (HIV) infection
* Contraindication or history of allergic reaction to one of the treatment components.
* Previous irradiation (external radiotherapy or brachytherapy) within 30 days prior to study treatment.
* Major surgery within 30 days prior to study treatment.
* Participation in another clinical trial within 30 days prior to study treatment.
* Concomitant systemic immunotherapy, chemotherapy, antitumor hormone therapy, targeted therapy or any experimental therapy.
* Active uncontrolled infection, peripheral neuropathy grade ≥ 2, acute or subacute bowel obstruction, history of inflammatory bowel disease, interstitial pneumonitis, respiratory failure, renal failure, dysphagia or any malabsorption condition.
* Symptomatic coronary heart disease or myocardial infarction in the past 6 months, congestive heart failure (NYHA class II), prior cerebrovascular accident.
* Uncontrolled hypertension (systolic blood pressure (BP) > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
* Proteinuria of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) ≥ grade 2 (i.e. urinary protein ≥ 1.0 g/24 hrs).
* Patients with current or anticipated need for strong Cytochrome P450 3A4 (CYP3A4) inhibitors or inducers.
* Pregnancy (or positive β-HCG dosage at inclusion), breast-feeding, or lack of effective contraception in male or female patients of reproductive potential.
* Other malignancies either currently active or in the last 5 years, except adequately treated in situ carcinoma of the cervix and basal or squamous cell skin carcinoma.
* Legal incapacity or physical, psychological or mental status interfering with the patient's ability to sign the informed consent or to terminate the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Limiting toxicity | up to 5 years
  To assess Limiting Toxicities during and within 6 weeks (2 cycles) after the beginning of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: DOMERGUE Jacques, Study Director — Institut régional du Cancer - Val d'Aurelle
Locations (1):
- Centre Val d'Aurelle, Montpellier, France

REFERENCES:
- [Derived] Blanc JF, Bouattour M, Gauthier L, Deshayes E, Guillemard S, Touchefeu Y, Portales F, Borg C, Harguem L, Guimbaud R, Mineur L, Ychou M, Mazard T, Assenat E. Regorafenib plus modified gemcitabine-oxaliplatin in patients with advanced biliary tract cancer. The randomized phase Ib/II BREGO study. Oncologist. 2025 Jun 4;30(6):oyaf080. doi: 10.1093/oncolo/oyaf080. PMID 40542585